CLINICAL TRIAL: NCT05135572
Title: What is the Relationship Between Tarsal Tunnel Syndrome and Foot Pain in Fibromyalgia Patients
Brief Title: Tarsal Tunnel Syndrome and Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MLeblebicier1
Record Dates: First submitted 2021-11-24; First posted 2021-11-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-11

CONDITIONS: Tarsal Tunnel Syndrome
Keywords: Tarsal Tunnel Syndrome, Fibromyalgia, Neuropathic pain, EMG
MeSH Terms: conditions — Tarsal Tunnel Syndrome; Fibromyalgia; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Fibromiyalgia patients with foot pain.
  Interventions: Diagnostic Test: Fibromiyalgia and foot pain
- study group (Experimental): Patients with foot pain
  Interventions: Diagnostic Test: Fibromiyalgia and foot pain

INTERVENTIONS:
Diagnostic Test: Fibromiyalgia and foot pain — Sensory and motor conduction studies will be performed in the lower extremities. Nerve conduction studies will be performed by another physician unaware of the patient's diagnosisFunctional status will be evaluated by using the Turkish version of the Fibromyalgia Impact Questionnaire (FIQ).Neuropathic Pain will be evalutaed by using the Turkish version of the Neuropathic Pain Questionnaire.
  Other Names: Patients with foot pain

SUMMARY:
Widespread pain is observed in patients diagnosed with fibromyalgia, and lower extremity and foot pain are also common. In our study, we aimed to evaluate the relationship between foot pain and tarsal tunnel syndrome in female patients diagnosed with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* Diagnosed with fibromyalgia according to ACR criteria

Exclusion Criteria:

* Have any severe mental or psychological disorder
* Have significant hearing and/or vision loss
* Presence of foot deformity, previous fracture, arthritis, tendon pathology that may cause foot pain detected in the physical examination of the foot and ankle joint.
* Presence of systemic inflammatory disease
* Having any systemic disease that may cause polyneuropathy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Electrodiagnostic studies | 15 minutes
  It is a neurological examination method based on the examination of the electrical potential of nerves and striated muscles.
Fibromyalgia Impact Questionnaire (FIQ) | 3 minutes
  This scale measures several patient characteristics over the past week: physical functioning, work status, depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being.The total FIQ score ranges from 0 to 100 and higher scores indicate severe effects of FMS. The minimal clinical important difference (MCID) for FIQ was reported to be minimum 14% or 8.1-point improvement
Neuropathic Pain Questionnaire. | 3 minutes
  This scala measures the type of pain, whether it has changed over time, and whether the pain is in one or more regions.This scala measures the type of pain, whether it has changed over time, and whether the pain is in one or more regions. It consists of 12 questions. Each question is scored between 0 and 100 points. It is multiplied by the coefficients determined for each question. All the resulting values are summed up, including fixed numbers. The result of the sum reflects the discriminant function score. Individuals with a score below 0 are predicted to have non-neuropathic pain, while those with a score of 0 or higher are predicted to have neuropathic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Scıence University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No